CLINICAL TRIAL: NCT01902043
Title: CoDiab-VD: a Population-based Cohort on Quality of Care of Patients With Diabetes in the Canton of Vaud (Switzerland)
Acronym: CoDiab-VD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: Service de la santé publique, Canton de Vaud (Unknown); Swiss National Science Foundation (Other); Foundation Swiss School of Public Healthplus (Unknown)
Responsible Party: Principal Investigator, Peytremann Bridevaux Isabelle, Professor, Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland
Other Study IDs: CoDiab-VD-151/11
Record Dates: First submitted 2013-07-09; First posted 2013-07-17 (Estimated); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; cohort study; quality of care; quality indicators, Health care; quality of Health Care; outcome and process assessment; health services research; chronic diseases prevention and management
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Diabetes, one of the most prevalent chronic disease (~ 9% worldwide), represents a major public health burden in terms of morbidity, disability and mortality. Caring for patients with diabetes requires effective collaboration between healthcare providers, teamwork, self-management education and use of evidence-based medicine. However, these processes of care are complex and often suboptimal. Improving quality of diabetes care is thus needed to reduce the health and societal burden of this disease.

In the canton of Vaud, a state in Switzerland with more than 700,000 inhabitants, a recent population-based study has shown that the prevalence of diabetes was around 7%. Data on the quality of diabetes care is scarce and quality of care data are still infrequently and unsystematically collected in Switzerland. In addition, when data are available, they focus on intermediate outcomes as well as clinical and biological cardiovascular risk factors. Population-based data on patient-reported outcomes are not considered.

In 2010, the Public Health Department of the canton of Vaud initiated the development of a regional diabetes program entitled "Programme cantonal Diabète" (PcD). It aimed both at decreasing the incidence of diabetes and improving care for patients with diabetes.

To tailor the program to the healthcare needs of patients and healthcare professionals involved in diabetes care, an exploratory study using qualitative methods was conducted in 2010. This was followed by a population-based survey conducted in fall 2011 and summer 2012. The objectives of the survey were to characterize patients with diabetes and assess the quality of the care they received. In addition, the results of the survey were used to help targeting unmet needs and possible areas of improvements, and constituted the patients' baseline measurement for the evaluation of the PcD.

The CoDiab-VD cohort emerged from that initial project; its specific objectives were 1) to follow over time the quality of diabetes care, 2) to explore topics that the PcD needed for its development, 3) to assess the impact of the PcD on the care of patients with diabetes, and 4) to evaluate the coverage of the PcD in the canton of Vaud.

DETAILED DESCRIPTION:
Diabetes, one of the most prevalent chronic disease (~ 9% worldwide), represents a major public health burden in terms of morbidity, disability and mortality. Caring for patients with diabetes requires effective collaboration between healthcare providers, teamwork, self-management education and use of evidence-based medicine. However, these processes of care are complex and often suboptimal. Improving quality of diabetes care is thus needed to reduce the health and societal burden of this disease.

In the canton of Vaud, a state in Switzerland with more than 700,000 inhabitants, a recent population-based study has shown that the prevalence of diabetes was around 7%. Data on the quality of diabetes care is scarce and quality of care data are still infrequently and unsystematically collected in Switzerland. In addition, when data are available, they focus on intermediate outcomes as well as clinical and biological cardiovascular risk factors. Population-based data on patient-reported outcomes are not considered.

In 2010, the Public Health Department of the canton of Vaud initiated the development of a regional diabetes program entitled "Programme cantonal Diabète" (PcD). It aimed both at decreasing the incidence of diabetes and improving care for patients with diabetes.

To tailor the program to the healthcare needs of patients and healthcare professionals involved in diabetes care, an exploratory study using qualitative methods was conducted in 2010. This was followed by a population-based survey conducted in fall 2011 and summer 2012. The objectives of the survey were to characterize patients with diabetes and assess the quality of the care they received. In addition, the results of the survey were used to help targeting unmet needs and possible areas of improvements, and constituted the patients' baseline measurement for the evaluation of the PcD.

The CoDiab-VD cohort emerged from that initial project; its specific objectives were 1) to follow over time the quality of diabetes care, 2) to explore topics that the PcD needed for its development, 3) to assess the impact of the PcD on the care of patients with diabetes, and 4) to evaluate the coverage of the PcD in the canton of Vaud.

Patients with diabetes were recruited by community-based pharmacies in the fall of 2011 and the summer of 2012. Participating community-based pharmacies, randomly contacted among those registered in the canton of Vaud, were asked to recruit non-institutionalized adult patients with diabetes (disease duration of at least 12 months), who were visiting the pharmacy with a prescription for oral antidiabetic drugs, insulin, glycemic strips or glucose meter.

At baseline, patients filled in a self-reported paper questionnaire that targeted the following areas:

* diabetes characteristics (type, disease duration, treatment, complications)
* receipt of diabetes care: recommended process of care indicators (such as annual eye examination by ophthalmologist, foot examination, microalbuminuria…) , and specific outcomes of care (such as HbA1C levels, generic and specific (health-related) quality of life (SF-12 and ADDQoL))
* congruence of care with the chronic care model (PACIC)
* healthcare utilization
* health behaviors (smoking and drinking habits, physical activity) and health status (comorbidities)
* self-management support (for example glycemic self-monitoring, self-efficacy, information level about diabetes)
* sociodemographic characteristics (age, gender, nationality, place of residence, education, employment, marital status, family size, family income, insurance status).

Participants were also asked to give the contact details of their family doctor and/or diabetologist. With the consent of the patients, treating physicians were contacted and were asked to fill a brief paper questionnaire requesting some clinical and laboratory data. Physicians were contacted in 2011, 2012 and 2014; physicians' follow-up was not repeated thereafter due to financial and logistic constraints.

Patients were contacted annually using paper follow-up questionnaires, consisting in a core set of questions similar to the baseline questionnaire. New questions were added and developed yearly according to the development and needs of the PcD. This allowed us to investigate these specific topics: diabetic foot in 2013; psychosocial outcomes related to diabetes and diabetes care in 2014; eyes and diabetes, as well as coordination and continuity of care in 2015; multimorbidity and needs for patient education in 2016; and pharmacy care in 2017.

A second recruitment, requested and financed by the funders, has been organized in 2017, in order to obtain a new population-based picture of diabetes in the canton of Vaud. It will allow 1) to compare data obtained at both recruitments, 2) to compare data obtained in 2017 from the second recruitment and from the annual follow-up of the first recruitment, and 3) to increase the number of patients with diabetes included in the CoDiab-VD cohort.

If requested by the PcD, additional follow-ups will take place in 2019 and in 2021.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus
* Disease ≥ 12 months
* Age ≥ 18 years
* Residing in the canton of Vaud, Switzerland, non-institutionalized
* Informed consent

Exclusion Criteria:

* Gestational diabetes mellitus
* Obvious cognitive impairment
* Not speaking or understanding French well enough

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-institutionalized adult patients with diabetes (≥18 years, type 1 or 2 diabetes, disease duration ≥12 months) who were visiting the pharmacy with a prescription for oral antidiabetic drugs, insulin, glycemic strips or glucose meter, at the time of the recruitment, are eligible for this study.
Sampling Method: Probability Sample
Enrollment: 1033 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Process of care indicators and the following outcomes of care: HbA1C, quality of life (QoL), Patient Assessment of Chronic Illness Care (PACIC) | Baseline and follow up once a year up to 10 years

OTHER OUTCOMES:
"Self-management support" measures (glycemic self-monitoring, participation in education classes/groups, self-efficacy, use of the diabetes passport) | Baseline and follow up once a year up to 10 years
Knowledge of and participation in the activities/projects of the Programme cantonal Diabète (PcD) | Baseline and follow up once a year up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Peytremann Bridevaux, Professor, Principal Investigator — Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland
Locations (1):
- Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Hagon-Traub I, Hirsiger P, Bovet P, Ruiz J, Peytremann-Bridevaux I, Noth C, Hauschild M. Programme cantonal Diabète, présentation du programme. Lausanne: Service de la Santé Publique du canton de Vaud; 2010. [http://www.vd.ch/fileadmin/user_upload/themes/sante_social/services_soins/Diabete/fichiers_pdf/Programme_cantonal.pdf]
- [Background] Casillas A, Iglesias K, Flatz A, Burnand B, Peytremann-Bridevaux I. No consistent association between processes-of-care and health-related quality of life among patients with diabetes: a missing link? BMJ Open Diabetes Res Care. 2015 Jan 10;3(1):e000042. doi: 10.1136/bmjdrc-2014-000042. eCollection 2015. PMID 25621176
- [Background] Collet TH, Taffe P, Bordet J, Burnand B, Peytremann-Bridevaux I. Reproducibility of diabetes quality of care indicators as reported by patients and physicians. Eur J Public Health. 2014 Dec;24(6):1004-9. doi: 10.1093/eurpub/cku011. Epub 2014 Feb 17. PMID 24534326
- [Background] Flatz A, Casillas A, Stringhini S, Zuercher E, Burnand B, Peytremann-Bridevaux I. Association between education and quality of diabetes care in Switzerland. Int J Gen Med. 2015 Feb 25;8:87-92. doi: 10.2147/IJGM.S77139. eCollection 2015. PMID 25759596
- [Background] Gijs E, Zuercher E, Henry V, Morin D, Bize R, Peytremann-Bridevaux I. Diabetes care: Comparison of patients' and healthcare professionals' assessment using the PACIC instrument. J Eval Clin Pract. 2017 Aug;23(4):803-811. doi: 10.1111/jep.12720. Epub 2017 Mar 2. PMID 28251768
- [Background] Iglesias K, Burnand B, Peytremann-Bridevaux I. PACIC Instrument: disentangling dimensions using published validation models. Int J Qual Health Care. 2014 Jun;26(3):250-60. doi: 10.1093/intqhc/mzu042. Epub 2014 Apr 15. PMID 24737833
- [Background] Rosselet PC, Zuercher E, Pasquier J, Burnand B, Peytremann-Bridevaux I. Impact of forgoing care because of costs on the quality of diabetes care: A three-year cohort study. Eur J Intern Med. 2017 Jun;41:e35-e37. doi: 10.1016/j.ejim.2017.03.007. Epub 2017 Mar 11. No abstract available. PMID 28292557
- [Background] Zuercher E, Diatta ID, Burnand B, Peytremann-Bridevaux I. Health literacy and quality of care of patients with diabetes: A cross-sectional analysis. Prim Care Diabetes. 2017 Jun;11(3):233-240. doi: 10.1016/j.pcd.2017.02.003. Epub 2017 Mar 11. PMID 28292571
- [Background] Konstantinidis L, Carron T, de Ancos E, Chinet L, Hagon-Traub I, Zuercher E, Peytremann-Bridevaux I. Awareness and practices regarding eye diseases among patients with diabetes: a cross sectional analysis of the CoDiab-VD cohort. BMC Endocr Disord. 2017 Sep 7;17(1):56. doi: 10.1186/s12902-017-0206-2. PMID 28882117
- [Background] Bawab N, Zuercher E, Carron T, Chinet L, Bugnon O, Berger J, Peytremann-Bridevaux I. Interest in and use of person-centred pharmacy services - a Swiss study of people with diabetes. BMC Health Serv Res. 2021 Mar 10;21(1):216. doi: 10.1186/s12913-021-06217-6. PMID 33691691
- [Result] Peytremann-Bridevaux I, Bordet J, Zuercher E, Burnand B. Caractéristiques des patients diabétiques vaudois et évaluation de leur prise en charge : Rapport final (Recrutements 2011 et 2012). Lausanne : Institut universitaire de médecine sociale et préventive, 2013. (Raisons de santé, 211). [http://www.iumsp.ch/Publications/pdf/rds211_fr.pdf]
- [Result] Peytremann-Bridevaux I, Bordet J, Burnand B. Diabetes care in Switzerland: good, but perfectible: a population-based cross-sectional survey. BMC Health Serv Res. 2013 Jun 25;13:232. doi: 10.1186/1472-6963-13-232. PMID 23800376
- [Result] Peytremann-Bridevaux I, Bordet J, Santschi V, Collet TH, Eggli M, Burnand B. Community-based pharmacies: an opportunity to recruit patients? Int J Public Health. 2013 Apr;58(2):319-22. doi: 10.1007/s00038-012-0383-8. Epub 2012 Jul 1. No abstract available. PMID 22752242
- [Result] Zuercher E, Bordet J, Burnand B, Peytremann-Bridevaux I. CoDiab-VD: protocol of a prospective population-based cohort study on diabetes care in Switzerland. BMC Health Serv Res. 2015 Aug 14;15:329. doi: 10.1186/s12913-015-0991-0. PMID 26272346
- [Result] Zuercher E, Casillas A, Hagon-Traub I, Bordet J, Burnand B, Peytremann-Bridevaux I. Baseline data of a population-based cohort of patients with diabetes in Switzerland (CoDiab-VD). Swiss Med Wkly. 2014 May 26;144:w13951. doi: 10.4414/smw.2014.13951. eCollection 2014. PMID 24863132
- [Derived] Kosinski C, Zuercher E, Carron T, Chevallereau J, Le Pogam MA, Storari C, Wojtusciszyn A, Peytremann-Bridevaux I. Self-reported perceptions of adults with diabetes regarding their care and health in the time of COVID-19 pandemic in a Swiss region: a cross-sectional study. Swiss Med Wkly. 2024 Dec 5;154:3578. doi: 10.57187/s.3578. PMID 39835917